CLINICAL TRIAL: NCT03636295
Title: Low INR to Minimize Bleeding With Mechanical Valves Trial
Acronym: LIMIT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Emilie Belley-Cote, Principal Investigator, Population Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5139
Record Dates: First submitted 2018-07-25; First posted 2018-08-17 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Bleeding Post-mechanical Valve Replacement; Thromboembolism Post-mechanical Valve Replacement
Keywords: Mechanical valve replacement; Vitamin K antagonist; INR targets; Bleeding; Thromboembolism
MeSH Terms: conditions — Hemorrhage; Thromboembolism | interventions — Warfarin

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, open-label, blinded end-point (PROBE) clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Reduced INR Target (Experimental): Warfarin therapy will be titrated to a target INR in the range of 1.5 to 2.5.
  Interventions: Drug: Warfarin
- Standard INR Target (Active Comparator): Warfarin therapy will be titrated to a "standard of care" target INR range.
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Warfarin — Participants in both arms will be on warfarin therapy post-mechanical valve replacement as is standard, but will have different INR target ranges.
  Other Names: Coumadin

SUMMARY:
This study evaluates the use of a lower INR target (1.5 to 2.5) in patients with a mechanical bileaflet heart valve in the aortic position. This study will inform physicians about whether a lower INR target will decrease the risk of bleeding or increase the risk of blood clot formation and stroke. These results have the potential to reduce the burden of bleeding in patients with a mechanical heart valve who require lifelong warfarin (Coumadin) treatment.

DETAILED DESCRIPTION:
Warfarin (Coumadin) is a blood thinner used to prevent blood clot formation in patients with mechanical heart valves. Blood clots can block blood flow to the brain, heart, or other parts of the body. Mechanical heart valves increases the risk of clot so patients with a mechanical heart valve must take warfarin to reduce their risk of stroke and other blood clot-related problems.

The degree to which warfarin 'works' varies from person to person, and so dosage is determined by measuring each person's response to the drug as an 'international normalized ratio' or INR. A patient with an INR over 1.0 has blood that takes longer to clot than average, and increasing INR values represent increasing time required for blood to clot. While an INR over 1.0 decreases clotting risk, it also increases bleeding risk. It is important to carefully balance these risks.

Specific INR targets have been recommended for patients with a mechanical heart valve, but these recommendations differ between scientific groups and are based on low quality evidence. Recent studies suggest that a lower INR target range than is currently recommended can be used safely. A laboratory study showed that warfarin effectively prevents blood clot formation on mechanical heart valves as long as the INR is 1.5 or above. Two moderately-sized clinical studies showed that an INR target range of 1.5-2.5 resulted in less bleeding than the usual higher target range without increasing blood clot formation or stroke in patients with a newer valve model. Whether we could use a lower INR target range for patients with a mechanical aortic valve remains controversial.

This study evaluates the use of a lower INR target (1.5 to 2.5) in patients with a mechanical bileaflet heart valve in the aortic position. This study will inform physicians about whether a lower INR target will decrease the risk of bleeding or increase the risk of blood clot formation and stroke. These results have the potential to reduce the burden of bleeding in patients with a mechanical heart valve who require lifelong warfarin (Coumadin) treatment.

ELIGIBILITY:
Inclusion criteria:

* Age is 18 or older at the time of enrolment
* Have had a bileaflet mechanical heart valve implant in the aortic position 3 or more months ago
* Written informed consent from either the patient or substitute decision maker

Exclusion criteria:

* Has a second implanted mechanical valve (any position)
* Lower boundary of planned INR range is less than 2.0
* Pregnant or expecting to become pregnant during the study follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2625 (Estimated)
Dates: Start 2019-09-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Thrombosis/thromboembolism | Through study completion, an expected mean of 2-3 years
  Number of patients who have at least one of the following: ischemic stroke, systemic thromboembolism, and valve thrombosis
Major bleeding | Through study completion, an expected mean of 2-3 years
  Number of patients that have bleeding that results in the following:
  1. Death and/or,
  2. Symptomatic bleeding in critical area or organ (e.g. intracranial, intraspinal, intraocular, retroperitoneal, intraarticular, pericardial, in a non-operated joint, or intramuscular with compartment syndrome) and/or,
  3. Bleeding that causes drop of hemoglobin level by 20 g/L or more, or that requires the transfusion of 2 or more units of packed red blood cells or whole blood

SECONDARY OUTCOMES:
All cause mortality | Through study completion, an expected mean of 2-3 years
  Selected rather than cardiovascular mortality, as cause-specific mortality is often difficult to ascertain or define in complex cardiovascular patients in whom multi-end-organ dysfunction may accompany cardiovascular decline.
All clinically important bleeding | Through study completion, an expected mean of 2-3 years
  Number of patients that experience all clinically important bleeding (major and minor)
Minor bleeding | Through study completion, an expected mean of 2-3 years
  Number of patients that experience a bleed that does not meet major bleeding criteria
All stroke | Through study completion, an expected mean of 2-3 years
  Number of patients that experience a strokes, including ischemic stroke, ischemic with secondary transformation, stroke of uncertain classification and hemorrhagic stroke
Ischemic stroke | Through study completion, an expected mean of 2-3 years
  Number of patients that experience an ischemic stroke, defined as focal brain infarction caused by an arterial (or rarely venous) obstruction and as documented by CT/MRI that is normal or shows an infarct in the clinicall expected area
Hemorrhagic stroke | Through study completion, an expected mean of 2-3 years
  Number of patients that experience a hemorrhagic stroke, defined as requiring neuroimaging or autopsy confirmation, and includes two subcategories: primary intracerebral hemorrhage and primary subarachnoid hemorrhage
Type 1, 2 or 3 myocardial infarction | Through study completion, an expected mean of 2-3 years
  Number of patients who experience a type 1, 2 or 3 myocardial infarction
Systemic thromboembolism | Through study completion, an expected mean of 2-3 years
  Number of patients who experience a systemic thromboembolism
Valve thrombosis | Through study completion, an expected mean of 2-3 years
  Number of patients who experience a valve thrombosis
Pulmonary embolism | Through study completion, an expected mean of 2-3 years
  Number of patients who experience a pulmonary embolism
Deep vein thrombosis | Through study completion, an expected mean of 2-3 years
  Number of patients who experience a deep vein thrombosis
New renal replacement therapy | Through study completion, an expected mean of 2-3 years
  Number of patients requiring new renal replacement therapy
Time in therapeutic range | Through study completion, an expected mean of 2-3 years
  The percentage of time the patient's INR was within the target range
Proportion of patients with extreme INR values (>4) | Through study completion, an expected mean of 2-3 years
  The proportion of patients with at least one reported INR value above 4

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Belley-Côté, MD, MSc, Principal Investigator — McMaster University
Locations (35):
- Belgium (4):
  - Ziekenhuis Oost-Limburg, Genk, Limburg
  - AZ Oostende, Ostend, West-Vlaanderen
  - Imelda Hospital, Keerbergen
  - Universitair Ziekenhuis Leuven, Leuven
- University of Botswana, at Princess Marina Hospital, Gaborone, Botswana
- Brazil (5):
  - Sociedade Hospitalar Angelina Caron, Campina Grande do Sul, Paraná
  - HEW Cardiologia LTDA, Joinville, Santa Catarina
  - InCor-HCFMUSP, Cerqueira César, São Paulo
  - Fundação Universitária de Cardiologia mantededora do Instituto de Cardiologia e Transplantes do Distrito Federal, Brasília
  - Dante Pazzanese Institute of Cardiology, São Paulo
- St. Elizabeth Catholic General Hospital, Kumbo, Cameroon
- Canada (5):
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - Hamilton General Hospital, Hamilton, Ontario
  - London Health Sciences Centre Research Inc., London, Ontario
  - The Ottawa Hospital Research Institute, Ottawa, Ontario
  - Jewish General Hospital, Montreal, Quebec
- Fuwai Hospital, CAMS & PUMC, Beijing, China
- Denmark (3):
  - Esbjerg & Grindsted Hospital - University Hospital of Southern Denmark, Esbjerg, Region Syddanmark
  - Southern Jutland Hospital, Aabenraa
  - Aarhus University Hospital, Aarhus
- Universitätsklinikum Jena, Jena, Germany
- Italy (2):
  - Città di Lecce Hospital, Lecce, Apulia
  - Azienda Ospedaliero Universitaria Policlinico Riuniti Foggia, Foggia
- Nepal (3):
  - Shahid Gangalal National Heart Centre, Kathmandu, Bagmati
  - Nobel Medical College and Teaching Hospital, Biratnagar, Koshi
  - BP Koirala Institute of Health Sciences, Dharān, Koshi
- Erasmus University Medical Centre, Rotterdam, Netherlands
- Shifa Clinical Research Center, Islamabad, Capital Territory, Pakistan
- Meshalkin National Medical Research Center, Novosibirsk, Russia
- King Faisal Specialist Hospital & Research Centre, Riyadh, Saudi Arabia
- Soonchunhyang University Gumi Hospital, Gumi, South Korea
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain
- United Kingdom (3):
  - Golden Jubilee National Hospital, Clydebank, Glasgow
  - Liverpool Heart & Chest Hospital, Liverpool
  - South Tees Hospitals NHS Foundation Trust of The James Cook University Hospital, Middlesbrough

IPD SHARING:
Plan to Share IPD: No
We will establish a plan for the full-scale study but there is no plan to make IPD available to other researchers.

REFERENCES:
- [Background] Puskas J, Gerdisch M, Nichols D, Quinn R, Anderson C, Rhenman B, Fermin L, McGrath M, Kong B, Hughes C, Sethi G, Wait M, Martin T, Graeve A; PROACT Investigators. Reduced anticoagulation after mechanical aortic valve replacement: interim results from the prospective randomized on-X valve anticoagulation clinical trial randomized Food and Drug Administration investigational device exemption trial. J Thorac Cardiovasc Surg. 2014 Apr;147(4):1202-1210; discussion 1210-1. doi: 10.1016/j.jtcvs.2014.01.004. Epub 2014 Jan 12. PMID 24512654
- [Background] Torella M, Torella D, Chiodini P, Franciulli M, Romano G, De Santo L, De Feo M, Amarelli C, Sasso FC, Salvatore T, Ellison GM, Indolfi C, Cotrufo M, Nappi G. LOWERing the INtensity of oral anticoaGulant Therapy in patients with bileaflet mechanical aortic valve replacement: results from the "LOWERING-IT" Trial. Am Heart J. 2010 Jul;160(1):171-8. doi: 10.1016/j.ahj.2010.05.005. PMID 20598989